CLINICAL TRIAL: NCT03838666
Title: Utilization of Autologous Mesenchymal Cells to Enhance Rotator Cuff Repair - a Prospective Non-randomized, Open-Label Study to Assess the Safety and the Efficacy
Brief Title: Utilization of AMSC to Enhance Rotator Cuff Repair - Safety and Efficacy
Acronym: AMSC-RC-001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Primary endpoint (safety) has been achieved
Sponsor: Bioinova, s.r.o. (Industry)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMSC-RC-001
Record Dates: First submitted 2019-01-14; First posted 2019-02-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspension of human autologous MSC 3P (Experimental): Patients will receive perioperative hAMSC (1.5 ml) treatment in order to accelerate the healing of the surgically repaired rotator cuff and increase the mechanical properties of the tendon.
  Interventions: Drug: Suspension of human autologous MSC 3P

INTERVENTIONS:
Drug: Suspension of human autologous MSC 3P — Single administration of the suspension of human autologous MSC 3P in 1.5 ml on the surface of the repaired rotator cuff tendon
  Other Names: hAMSC

SUMMARY:
Subjects received perioperative hAMSC treatment in order to accelerate the healing of the surgically repaired rotator cuff and increase the mechanical properties of the tendon, according to inclusion and exclusion criteria (see below). Each patient will undergo post-operative follow-up at 6 weeks, 6 months and 12 months after the surgery. This will include a visual analogue score for pain (VAS), a questionnaire for the subjective Constant shoulder score, and the subjective questions of the University of California (UCLA) score. Preoperative and postoperative MRI at 12 months will be done to evaluate the quality of the rotator cuff repair.

DETAILED DESCRIPTION:
Eligible patients will undergo an arthroscopic rotator cuff repair augmented by mesenchymal stem cells (MSCs). The primary objective of the trial is to assess the safety and tolerability of autologous mesenchymal stem cells treatment applied during arthroscopic rotator cuff repair.

The condition of the patient will be monitored throughout the study. At each visit, adverse events (AEs) will be elicited using a standard non-leading questions. In addition, any signs or symptoms will be observed. All AEs will be collected as:

* patient's positive response to questions about their health
* symptoms spontaneously reported by the patient
* clinically relevant changes and abnormalities observed by the Investigator (e.g. local and systemic tolerability, clinically significant laboratory measurements confirmed by repeated measurement, results of physical examinations).

Clinical improvement will be measured by clinical outcome scores (Constant shoulder score and UCLA Shoulder rating scale) at 6 weeks, 6 months and 1 year after the surgery. MRI (Magnetic Resonance Imaging) findings made preoperatively and at 12 months (1 year) after operation will be evaluated.

During the indication visit, patient's history will be taken and preoperative MRI evaluated. Written consent form will be collected from the patient after detailed education of the patient by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. males or females between 40 and 65 years of age,
2. written informed consent obtained,
3. complete unilateral rotator cuff tear on pre-operative clinical and imaging findings,
4. elected to undergo an arthroscopic repair of their rotator cuff tear,
5. agreed to wear a dedicated brace for four weeks post-operatively,
6. minimum pre-operative hemoglobin of 11.0 g/dl or more
7. pre-operative platelet count greater than 150 000 / 1 mm3

Exclusion Criteria:

1. a tear involving the subscapularis or biceps tendons,
2. a previous rotator cuff repair,
3. moderate-to-severe osteoarthritis of the glenohumeral joint,
4. loss of passive elevation in any direction when compared to the contralateral shoulder,
5. fatty infiltration greater than 50 % of the cross-sectional area of supraspinatus or infraspinatus assessed on the most lateral image on which the scapular spine is in contact with the scapular body,
6. a massive tear with a contracted immobile cuff confirmed in operation,
7. an active infection, osteomyelitis or sepsis or distant infections which may spread to the site of operation,
8. other diseases which may have limit follow-up (immunocompromising, hepatitis, active tuberculosis, neoplastic diseases, septic arthritis),
9. osteomalacia or other metabolic bone disorders which may impair bone or soft tissue function,
10. vascular insufficiency, muscular atrophy or neuromuscular diseases of the affected arm,
11. haemato/oncological diseases,
12. pregnant or lactating women,
13. alcohol or drug abusers,
14. patients on corticosteroids, immunosuppressants or anticoagulant therapy,
15. women of childbearing potential not using effective contraception (established oral contraception, intrauterine device, ligation of the uterine tube) including proven contraceptive measures taken by their sexual partners,
16. fertile men not using proven contraceptive measures including effective contraception of their partners (established oral contraception, intrauterine device, ligation of the uterine tube).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2015-11-18 (Actual)

PRIMARY OUTCOMES:
Safety: To assess the occurrence of adverse events of treatment by hAMSC - systemic reactions. | 1 year
  Safety and tolerability of hAMSC treatment applied during the surgical rotator cuff repair will be recorded - systemic reactions including allergic reaction or sepsis at Visits I through VI.
Safety: To assess the occurrence of adverse events of treatment by autologous mesenchymal stem cells - local reactions. | 1 year
  Safety and tolerability of autologous mesenchymal stem cells treatment applied during the surgical rotator cuff repair will be recorded - local reactions including pain, bleeding, local infection at Visits I through VI.

SECONDARY OUTCOMES:
Efficacy: To evaluate the effect of hAMSCs applied during arthroscopic rotator cuff repair - Visual Analogue Score (VAS) | 1 year
  The efficacy analysis will be evaluated by comparing pre- and post-treatment rotator cuff function measured by changes in Visual Analogue Score (VAS) (meter-shaped scale; in mm) at Visits II, IV, V, and VI.
  VAS is a self-report measure consisting simply of a 10 centimeter line with a statement at each end representing one extreme of the dimension being measured (most often intensity of pain). The respondent gives their indication with a pen mark on the line corresponding to their answer, e.g. the present pain level.
Efficacy: To evaluate the effect of hAMSCs applied during arthroscopic rotator cuff repair - Constant Shoulder Score | 1 year
  The secondary efficacy analysis will be evaluated by comparing pre- and post-treatment rotator cuff function by changes in Constant Shoulder Score (points) at Visits II, IV, V, and VI.
  Measurements: Pain, Activities of daily living, Range of movement (forward flexion, abduction, external rotation, internal rotation), Power.
  Less points (out of 100) means more severe condition.
Efficacy: To evaluate the effect of hAMSCs applied during arthroscopic rotator cuff repair - UCLA Shoulder Rating Score | 1 year
  The secondary efficacy analysis will be evaluated by comparing pre- and post-treatment rotator cuff function by changes in UCLA Shoulder Rating Score (points) at Visits II, IV, V, and VI.
  Measurements: Pain, Function, Active forward flexion, Strength of forward flexion (manual muscle-testing), Satisfaction of patient.
  Less points (out of 35) means more severe condition.
Efficacy: To evaluate the effect of hAMSCs applied during arthroscopic rotator cuff repair - MRI imaging - Continuation / discontinuation of the rotator cuff | 1 year
  The secondary efficacy analysis will be evaluated by comparing pre- and post-treatment rotator cuff function which measured by MRI imaging (preoperative and at Visit VI) to evaluate the quality of the rotator cuff repair.
  Following finding will be recorded:
  * Continuation / discontinuation of the rotator cuff
  * preoperatively - confirmation of complete unilateral rotator cuff tear
  * 1 year after the treatment (Visit VI) - the quality and extent of rotator cuff repair - no recovery/partial recovery/full recovery
Efficacy: To evaluate the effect of hAMSCs applied during arthroscopic rotator cuff repair - MRI imaging - Fatty degeneration | 1 year
  The secondary efficacy analysis will be evaluated by comparing pre- and post-treatment rotator cuff function which measured by MRI imaging (preoperative and at Visit VI) to evaluate the quality of the rotator cuff repair.
  Following finding will be recorded:
  - Amount of fatty degeneration - percentage of fatty infiltration of the cross sectional area of supraspinatus or infraspinatus assessed on the most lateral image on which the scapular spine is in contact with the scapular body,

CONTACTS AND LOCATIONS:
Overall Officials: Petr Lesny, MD, Study Chair — Bioinova, s.r.o.

IPD SHARING:
Plan to Share IPD: No
The data has been published